CLINICAL TRIAL: NCT07054255
Title: Bioequivalence and Safety Study of Ranolazine Extended-release Tablets in Healthy Chinese Subjects Under Fasting and Fed Conditions: A Randomized, Open-label, Single-dose, Cross-over Study
Brief Title: Bioequivalence Study of Ranolazine Extended-release Tablets in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HSK-63-BE-2020
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test formulation (Experimental): Ranolazine sustained-release tablets, specification: 500 mg, Haisco Pharmaceutical Co., Ltd.
  Interventions: Drug: Test formulation (Ranolazine extended-release tablets)
- Reference formulation (Experimental): Ranolazine sustained-release tablets (Ranexa®), specification: 500 mg, Gilead Sciences, Inc.
  Interventions: Drug: Reference formulation (Ranolazine extended-release tablets)

INTERVENTIONS:
Drug: Test formulation (Ranolazine extended-release tablets) — A single oral dose of 500 mg, taken with 240mL of water
  Arms: Test formulation
Drug: Reference formulation (Ranolazine extended-release tablets) — A single oral dose of 500 mg, taken with 240mL of water
  Arms: Reference formulation

SUMMARY:
The present study was conducted with the objective of comparing the bioequivalence and safety of a single dose of ranolazine extended-release tablets (Test product) manufactured by Haisco Pharmaceutical Group Co., Ltd. with those of the reference product (Ranexa®, Gilead Sciences, Inc.) in Chinese healthy subjects under fasting and fed conditions

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged 18 or older, both male and female, with an appropriate gender ratio;
2. Female subjects weight ≥ 45.0 kg and male subjects weight ≥ 50.0 kg, and BMI of 19 to 26 kg/m^2(inclusive);
3. Subjects who have no plans to conceive or donate sperm/eggs during the trial period until 3 months after the end of the trial and voluntarily adopt effective physical contraception measures.
4. Prior to the trial, a detailed understanding of the nature, significance, potential benefits, potential inconvenience, risks, and discomfort of the trial was obtained, and the subjects voluntarily participated in the clinical trial. The subject was able to communicate well with the researchers, comply with the requirements of the entire study, and signed a written informed consent form.

Exclusion Criteria:

1. Subjects who are known to be allergic to the investigational drug component Ranolazine (including excipients) or similar substances, or those with an allergic constitution (such as allergies to two or more drugs, food, or pollen) (consultation);
2. Subjects with a history of chronic or severe diseases or existing systemic diseases that may affect the research results, including those related to the blood system, circulatory system, digestive system, urinary system, respiratory system, nervous system, immune system, endocrine system, mental disorders, metabolic disorders, or any other conditions that may affect the research results (consultation);
3. Subjects who have undergone major surgery or suffered severe trauma within the first 3 months (90 days) of screening, or who have undergone surgery that may significantly affect the in vivo process or safety evaluation of the study drug (consultation);
4. Received vaccination within one month (30 days) before screening(consultation);
5. Used any prescription medication (such as antihypertensive drugs) within 1 month (30 days) before screening, or used any over-the-counter medication (vitamins, herbal medicines) within 2 weeks before screening (consultation);
6. Subjects who have participated in and used any clinical trial drug or medical device within 3 months (90 days) before the first administration, or those who plan to participate in other clinical trials during this study (consultation);
7. Subjects who regularly drink alcohol within one month (30 days) before screening (drinking alcohol ≥ 3 times a week, and drinking 50 ° Baijiu ≥ 100 mL each time on average), or cannot abstain from alcohol during the test, or the alcohol breath test result is>0.000mg/mL (consultation, examination);
8. Subjects who have been addicted to smoking (more than 5 cigarettes per day or an equivalent amount of tobacco) for the past 3 months (90 days) prior to screening or who cannot stop using any tobacco products during the trial period (consultation);
9. Subjects who have lost blood/donated more than 400 mL (excluding physiological blood loss in females) within 2 months (60 days) prior to screening, or who have received blood transfusions/used blood products, or who plan to donate blood within 1 month (30 days) after the end of the trial (consultation);
10. On a daily within 2 weeks prior to screening,consuming excessive amounts of foods that affect metabolism, such as grapefruit or beverages containing grapefruit; Consuming excessive amounts of tea, coffee, chocolate, cola, or foods/beverages containing their main ingredients every day (averaging 8 or more cups per day, 200 mL per cup); Diets rich in xanthine, flavonoids, and other components (consultation);
11. Within 48 hours before the first administration, consume grapefruit or beverages containing grapefruit; Consuming tea, coffee, chocolate, cola, or foods/beverages containing their main ingredients; Consuming a diet rich in xanthine, flavonoids, and other components; Or those who engage in vigorous exercise (consultation);
12. Subjects with a history of drug abuse or positive results in urine drug abuse screening (consultation, examination);
13. Any positive subject in screening period virus serum blood examination (hepatitis B surface antigen, hepatitis C antibody, HIV antigen antibody, Treponema pallidum antibody);
14. During the screening period, if the physical examination, vital signs, electrocardiogram or laboratory test results are judged by clinical doctors to be abnormal and clinically significant, or if the QT interval is prolonged (female QT>440 ms or male QT>420 ms), or if fasting blood glucose exceeds the upper limit of normal values (examination);
15. Pregnant or lactating women, or those who test positive for pregnancy (consultation, examination);
16. Subjects who are prone to diarrhea, nausea, vomiting, bloating, or other gastrointestinal discomfort after drinking milk or dairy products, or who are prone to dizziness, headache, constipation, and nausea on a regular basis (consultation);
17. Subjects with a history of needle dizziness, blood dizziness, or intolerance to venipuncture blood collection (for consultation and examination);
18. Subjects with difficulty swallowing tablets/capsules (consultation);
19. Subjects with special dietary requirements (such as vegetarians) or those who cannot adhere to a uniform diet during the trial period (consultation);
20. Subjects who may not be able to cooperate with the completion of the study for other reasons, or the investigator may determine that they are not suitable for inclusion;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-09-06 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Cmax | From the start of administration to 48 hours post-dose
  The pharmacokinetic parameters of Ranolazine in plasma
AUC(0-t) | From the start of administration to 48 hours post-dose
  The pharmacokinetic parameters of Ranolazine in plasma
AUC(0-∞) | From the start of administration to 48 hours post-dose
  The pharmacokinetic parameters of Ranolazine in plasma

SECONDARY OUTCOMES:
AEs | From the time of signing ICF to the end of follow-up，up to 10 days
  The incidence and severity of AEs

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Chen X, Li Y, Ma G. Bioequivalence and Safety Study of Ranolazine Extended-Release Tablets in Chinese Healthy Subjects Under Fasting and Fed Conditions: A Randomized, Open-Label, Single-Dose, Cross-Over, Comparative Pharmacokinetic Study. Clin Ther. 2026 Jan;48(1):88-94. doi: 10.1016/j.clinthera.2025.11.002. Epub 2025 Nov 25. PMID 41298182